CLINICAL TRIAL: NCT05140512
Title: A Randomized, Open-label and Parallel Phase I Study to Compare Pharmacokinetics, Pharmacodynamics and Safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01005) and ZOLADEX® Following Multiple Administration in Patients With Prostate Cancer
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of LY01005 in Patients With Prostate Cancer Compared to ZOLADEX®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01005/CT-CHN-104
Record Dates: First submitted 2021-11-03; First posted 2021-12-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; LY01005; PK/PD; Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01005 3.6 mg (Experimental): Intramuscular injections of LY01005 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: LY01005
- ZOLADEX® 3.6 mg (Active Comparator): Subcutaneous injections of ZOLADEX® 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: ZOLADEX® 3.6 mg

INTERVENTIONS:
Drug: LY01005 — LY01005 was administered as 3 intramuscular (IM) injections, 28 days apart. As concomitant medications, Casodex® (50 mg/day) was orally administered during the whole study period.
  Other Names: Goserelin Acetate Sustained-Release Microspheres for Injection
  Arms: LY01005 3.6 mg
Drug: ZOLADEX® 3.6 mg — ZOLADEX® was administered as 3 Subcutaneous (SC) injections, 28 days apart. As concomitant medications, Casodex® (50 mg/day) was orally administered during the whole study period.
  Other Names: Goserelin Acetate Implant 3.6 mg
  Arms: ZOLADEX® 3.6 mg

SUMMARY:
This is a randomized, open-label and parallel phase I study to compare pharmacokinetics (PK), pharmacodynamics (PD) and safety of goserelin acetate sustained-release microspheres for injection (LY01005) and ZOLADEX® following multiple administration in patients with prostate cancer.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled phase I trial. A total of 23 patients with locally advanced or metastatic prostate cancer who were suitable for endocrine therapy were enrolled into the screening period from D-21 to D-10 (±3d) before administration. Eligible subjects were treated with bicalutamide tablets (Casodex®, 50 mg/day) from D-10 (± 3d) to the end of the trial and randomized in a 1:1 ratio to receive LY01005 3.6 mg or ZOLADEX ® 3.6 mg after completion of pretreatment. All subjects were administered once every 28 days for three doses. Blood samples were collected at the specified time points in the trial protocol to detect PK parameters of goserelin, and PD parameters (serum testosterone, LH and FSH). Safety evaluation (including vital signs, physical examination, laboratory tests, 12 ECG, adverse events, etc.) was conducted as required in the protocol. This study aimed to compare PK/PD and safety of LY01005 and ZOLADEX® in patients with locally advanced or metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patients with locally advanced or metastatic prostate cancer suitable for endocrine therapy, including those who are suitable for endocrine therapy (such as patients with biochemical recurrence after adjuvant endocrine therapy and radical therapy) following radical therapy.
* Serum testosterone level ≥ 150 ng/dL (1.50 ng/mL or 5.2 nmol/L) at the screening visit.
* Life expectancy of at least 9 months.
* ECOG score of ≤ 2.
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelet count ≥ 90 x 10^9/L, white blood cell count ≥ 3 x 10^9/L, hemoglobin ≥ 90 g/L, total bilirubin (TBIL) ≤ 1.5×ULN, ALT and AST ≤ 2.5×ULN (or ≤ 5.0×ULN for patients with liver metastases), and Creatinine clearance ≥50 mL/min at the screening visit.
* Subjects of childbearing potential must agree to use a reliable method of contraception with their female sexual partners during the study period and at least 3 months after the last administration.
* Patients who voluntarily sign an IRB-approved informed consent form before any trial-related activities, are willing to abide by the restrictions of the study, and complete the prescribed examinations.

Exclusion Criteria:

* Patients with prostate cancer who receive previous or ongoing endocrine therapy (surgical castration or other endocrine therapy including GnRH receptor agonists, GnRH receptor antagonists, anti-androgens, estrogens, megestrol acetate, etc.), except for patients with prostate cancer undergoing prostatectomy, radiotherapy or cryotherapy who have received neoadjuvant/adjuvant endocrine therapy for no more than 6 months and discontinued the above therapy more than 6 months before screening.
* Patients with confirmed or suspected hormone-resistant prostate cancer.
* Patients who have received prostatic surgery within 4 weeks prior to the first dose, or plan to receive major surgical treatment during the trial.
* Patients who have previously received hypophysectomy or adrenalectomy, or who have pituitary lesions or adrenal dysfunction.
* History of severe asthma, anaphylaxis, or severe urticaria and/or angioedema.
* Other cancer diseases diagnosed within 5 years before the screening visit, except for surgically removed basal or squamous cell carcinoma of the skin.
* History of the following medical histories within 6 months prior to the screening visit: stroke, transient ischemic attack (TIA), myocardial infarction, unstable angina, coronary revascularization, New York Heart Association (NYHA) class ≥ II cardiac insufficiency, severe unstable arrhythmia.
* Hypertensive patients with poor blood pressure control (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg at the screening visit).
* Patients with type 1 diabetes or type 2 diabetes with poor glycemic control (glycosylated hemoglobin > 8% at the screening visit).
* Patients who have received treatment with 5-α reductase inhibitors (finasteride, dutasteride, enalidomide, epristeride, etc.) within 4 weeks before the first dose.
* Has previously received goserelin.
* Is receiving coumarin anticoagulants at the screening visit.
* Has congenital long QT syndrome or QT/QTc interval prolongation (QTc ≥ 450 ms) at the screening visit; Or has received drugs that may prolong QT/QTc interval at the screening visit.
* Known to be allergic to the active ingredients or any excipients of GnRH agonists or bicalutamide.
* Patients who are seropositive for hepatitis B surface antigen (HBsAg), and must meet the following 2 conditions at the same time: 1. HBV DNA level: HBeAg-positive patients, HBV DNA ≥ 20,000 IU/ml [equivalent to 10^5 copies/mL]; HBeAg-negative patients, HBV DNA ≥ 2,000 IU/ml [equivalent to 10^4 copies/mL]; 2. ALT ≥ 2 x ULN); Patients who are seropositive for human immunodeficiency virus (HIV) antibody.
* Alcoholics or drug abusers. Alcoholics are defined as drinking more than 14 units of alcohol per week within 3 months prior to the screening visit (1 unit = 350 mL beer, or 45 mL liquor, or 150 mL wine).
* Has participated in any clinical trials of investigational drugs or medical devices, and discontinued within 1 month or 5 half-lives of the corresponding drug before the screening visit, whichever is longer.
* Other conditions considered unsuitable for enrollment by the investigator (such as spinal cord compression due to prostate cancer metastatic lesions of pyramid, pulmonary interstitial disease or other serious diseases).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Plasma concentration of goserelin over time. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Cmax. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Ctrough. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: AUC0-t. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: AUC0-∞. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Tmax. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: T1/2. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Vz/F. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: Cl/F. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: MRT0-∞. | from baseline to Day 85
Pharmacokinetic Profile of LY01005 versus ZoLADEX®: accumulation of goserelin. | from baseline to Day 85

SECONDARY OUTCOMES:
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: AUEC of serum testosterone. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: Emax of serum testosterone. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: TEmax of serum testosterone. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: AUEC of serum LH. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: Emax of serum LH. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: TEmax of serum LH. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: AUEC of serum FSH. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: Emax of serum FSH. | from baseline to Day 85
Pharmacodynamic Profile of LY01005 versus ZoLADEX®: TEmax of serum FSH. | from baseline to Day 85
The percentage of subjects with serum testosterone ≤50 ng/dL (1.735 nmol/L) on Day 29 after the first dose. | Day 29 after the first dose
The cumulative percentage of subjects with the maintenance of serum testosterone ≤50 ng/dL (1.735 nmol/L) from Day 29 to Day 85. | from Day 29 to Day 85
Significant Castration Rate. | from Day 29 to Day 85
  The percentage of subjects with serum testosterone ≤20 ng/dL (0.7 nmol/L) on Day 29 after the first dose, and the cumulative percentage of subjects with the maintenance of serum testosterone ≤20 ng/dL (0.7 nmol/L) from Day 29 to Day 85.
The percentage of subjects with serum testosterone > 50 ng/dL on 1 hour, 4 hours, Day 3 and Day 7 after the second dose and the third dose. | 1 hour, 4 hours, Day 3 and Day 7 after the second dose and the third dose
Percentage changes compared to baseline in serum FSH level after each administration. | Day 29, Day 57 and Day 85
Percentage changes compared to baseline in serum LH level after each administration. | Day 29, Day 57 and Day 85
Adverse events throughout the study. | up to Day 85

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No